CLINICAL TRIAL: NCT05661058
Title: MAPping Sedentary Behaviour (MAPS-B) in Older Adults: A Mix-methods Longitudinal Study
Brief Title: Mapping Sedentary Behaviour in Older Adults Who Are Frail
Acronym: MAPS-B
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Isabel Rodrigues (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Isabel Rodrigues, Postdoctoral fellow, McMaster University
Organization: McMaster University (Other)
Other Study IDs: MAPSB
Record Dates: First submitted 2022-12-06; First posted 2022-12-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Frailty
Keywords: Sedentary behaviour; Frailty; Falls; Old adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total number of participants: As this is not an intervention study, the investigators only have one group which the investigators will follow at two-time points to map the context of sedentary behaviour.

SUMMARY:
The purpose of this study is to map the context of sedentary behaviour among older adults who are frail. This study uses a unique combination of objective and self-report measures to assess context. The investigators will also hold focus groups to understand which behaviours can be modified and conduct an analysis to understand which types of behaviours are associated with negative health outcomes.

DETAILED DESCRIPTION:
Older adults who are frail are potentially the population that might benefit the most from a reduction in sedentary time as they are the most sedentary group and have the highest chronic disease burden. However, there is a dearth of evidence on effective interventions to reduce sedentary behaviour or total sedentary time in older adults, especially among individuals that are frail. Previous studies focused on reducing total sedentary time, while other studies aimed to increase physical activity levels with the assumption that sedentary time will be reallocated to physical activity. But, to date, such interventions have not been effective at reducing total sedentary behaviour time in older adults. Previous studies to reduce sedentary time and behaviour in older adults may not be effective because there is no research on the context of sedentary behaviour, about when and where to intervene, and which specific sedentary behaviours should be targeted. Almost all studies in older adults have assessed total sedentary time, which does not provide enough information to understand the context of sedentary behaviours. The main reason to understand context is because not all sedentary behaviours should be modified as some cognitively engaging sedentary behaviours (e.g., reading, socializing) appear to benefit health, while time spent in more passive activities may be detrimental. Therefore, the goal should not be to reduce total sedentary time, but rather identify sedentary behaviours that may be detrimental to the health of older adults who are frail.

Before we can develop an intervention to reduce sedentary behaviour among older adults, we must first assess the context of sedentary behaviour. Context is defined as the purpose of the sedentary behaviours, the location where the behaviours occur, the posture of the behaviours (e.g., lying, sitting), social context (e.g., alone or with others), and time of day the behaviours occur. The purpose of this study was to assess the feasibility of measuring the context of sedentary behaviour among older adults who are frail. We defined feasibility using recruitment, retention, and refusal rates (process) and the feasibility resource (i.e., can the tools capture context and are participants willing to use the tools). Our criteria for success were to recruit 20 participants within two months, 85% retention, and 20% refusal. Our secondary objectives are: 1) to determine the context of using objective and subjective measures to assess sedentary behaviours among older adults who are frail; 2) to identify which types of sedentary behaviours can be modified and when and where to intervene; and 3) to conduct an exploratory analysis to determine the association of certain types of sedentary behaviours on health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years and older;
2. Categorizes as frail on the FRAIL scale ≥ 3 of 5;
3. Lives in the Greater Hamilton Area (GHA)
4. Speaks English or can attend with a translator.

Exclusion Criteria:

1. Requires a wheelchair at least 55% of the awake day; needs to sit for long periods of time due to a medical condition; or not independently mobile (i.e., requires assistance from another individual to ambulate);
2. Has travel plans or other commitments that means missing >30% of the rollout study period;
3. Unable to follow two-step instructions.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The investigators aim to recruit 20 participants (65 years and older) living with frailty. The investigators will recruit males and females as gender may influence sedentary behaviour through socially constructed norms and roles and can be affected by differential access to resources, opportunities, and power. The investigators are collaborating with geriatricians at Hamilton Health Sciences to recruit participants. The physician will inform eligible participants of the study and provide participants with a number to contact the research assistant. The research assistant will speak with interested participants to confirm eligibility and enroll them in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility process and resources | Two months
  The purpose of this study was to assess the feasibility of measuring the context of sedentary behaviour among older adults who are frail. We defined feasibility using recruitment, retention, and refusal rates (process feasibility) and the feasibility resource (i.e., can the tools capture context and are participants willing to use the tools). Our criteria for success for process feasibility were to recruit 20 participants within two-months with 85% retention by end of study, and a 20% refusal rate.

SECONDARY OUTCOMES:
Focus group (Winter) | 1 day
  The investigators will hold focus groups in groups of 5 participants or less after the winter collection periods to mitigate recall bias. The investigators will use semi-structured interviews to guide the focus group. Transcripts will be transcribed verbatim and analyzed in NVivo using codebook reliability thematic analysis
Regression analysis (Winter) | 7 consecutive days
  The investigators will conduct an exploratory analysis of secondary outcomes using multiple linear regression in SPSS Statistics version 27 (IBM Corp, Armonk, New York, USA). The independent variable will be the most common sequences of sedentary behaviour during the Winter period, and the dependent variable will be the secondary health outcomes (e.g., frailty level, cognitive status). The covariates will include variables from PROGRESS (i.e., age and sex).
Focus group (Spring) | 1 day
  The investigators will hold focus groups in groups of 5 participants or less after the spring collection periods to mitigate recall bias. The investigators will use semi-structured interviews to guide the focus group. Transcripts will be transcribed verbatim and analyzed in NVivo using codebook reliability thematic analysis
Regression analysis (Spring) | 3 consecutive days (2 weekdays and 1 weekend)
  The investigators will conduct an exploratory analysis of secondary outcomes using multiple linear regression in SPSS Statistics version 27 (IBM Corp, Armonk, New York, USA). The independent variable will be the most common sequences of sedentary behaviour during the Spring period, and the dependent variable will be the secondary health outcomes (e.g., frailty level, cognitive status). The covariates will include variables from PROGRESS (i.e., age and sex).
Context of sedentary behaviour (Winter) | Weekday #1
  Data analyses from the activPAL4TM and indoor positioning system and participants' diaries will be mapped to the Sedentary behaviour International Taxonomy (SIT) using classification scheme content analysis. SIT is a framework developed to help researchers understand the context and determinants of sedentary behaviours. The investigators will post process the data from the indoor positioning system in 15-minute intervals.
Context of sedentary behaviour (Winter) | Weekday #2
  Data analyses from the activPAL4TM and indoor positioning system and participants' diaries will be mapped to the Sedentary behaviour International Taxonomy (SIT) using classification scheme content analysis. SIT is a framework developed to help researchers understand the context and determinants of sedentary behaviours. The investigators will post process the data from the indoor positioning system in 15-minute intervals.
Context of sedentary behaviour (Winter) | Weekend #1
  Data analyses from the activPAL4TM and indoor positioning system and participants' diaries will be mapped to the Sedentary behaviour International Taxonomy (SIT) using classification scheme content analysis. SIT is a framework developed to help researchers understand the context and determinants of sedentary behaviours. The investigators will post process the data from the indoor positioning system in 15-minute intervals.
Context of sedentary behaviour (Spring) | Weekday #1
  Data analyses from the activPAL4TM and indoor positioning system and participants' diaries will be mapped to the Sedentary behaviour International Taxonomy (SIT) using classification scheme content analysis. SIT is a framework developed to help researchers understand the context and determinants of sedentary behaviours. The investigators will post process the data from the indoor positioning system in 15-minute intervals.
Context of sedentary behaviour (Spring) | Weekday #2
  Data analyses from the activPAL4TM and indoor positioning system and participants' diaries will be mapped to the Sedentary behaviour International Taxonomy (SIT) using classification scheme content analysis. SIT is a framework developed to help researchers understand the context and determinants of sedentary behaviours. The investigators will post process the data from the indoor positioning system in 15-minute intervals.
Context of sedentary behaviour (Spring) | Weekend #1
  Data analyses from the activPAL4TM and indoor positioning system and participants' diaries will be mapped to the Sedentary behaviour International Taxonomy (SIT) using classification scheme content analysis. SIT is a framework developed to help researchers understand the context and determinants of sedentary behaviours. The investigators will post process the data from the indoor positioning system in 15-minute intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walston J, Hadley EC, Ferrucci L, Guralnik JM, Newman AB, Studenski SA, Ershler WB, Harris T, Fried LP. Research agenda for frailty in older adults: toward a better understanding of physiology and etiology: summary from the American Geriatrics Society/National Institute on Aging Research Conference on Frailty in Older Adults. J Am Geriatr Soc. 2006 Jun;54(6):991-1001. doi: 10.1111/j.1532-5415.2006.00745.x. PMID 16776798
- [Result] Abellan van Kan G, Rolland YM, Morley JE, Vellas B. Frailty: toward a clinical definition. J Am Med Dir Assoc. 2008 Feb;9(2):71-2. doi: 10.1016/j.jamda.2007.11.005. No abstract available. PMID 18261696
- [Result] Bunt S, Steverink N, Olthof J, van der Schans CP, Hobbelen JSM. Social frailty in older adults: a scoping review. Eur J Ageing. 2017 Jan 31;14(3):323-334. doi: 10.1007/s10433-017-0414-7. eCollection 2017 Sep. PMID 28936141
- [Result] Gale CR, Westbury L, Cooper C. Social isolation and loneliness as risk factors for the progression of frailty: the English Longitudinal Study of Ageing. Age Ageing. 2018 May 1;47(3):392-397. doi: 10.1093/ageing/afx188. PMID 29309502
- [Result] Petrusevski C, Choo S, Wilson M, MacDermid J, Richardson J. Interventions to address sedentary behaviour for older adults: a scoping review. Disabil Rehabil. 2021 Oct;43(21):3090-3101. doi: 10.1080/09638288.2020.1725156. Epub 2020 Feb 14. PMID 32058808
- [Result] Chastin S, Gardiner PA, Harvey JA, Leask CF, Jerez-Roig J, Rosenberg D, Ashe MC, Helbostad JL, Skelton DA. Interventions for reducing sedentary behaviour in community-dwelling older adults. Cochrane Database Syst Rev. 2021 Jun 25;6(6):CD012784. doi: 10.1002/14651858.CD012784.pub2. PMID 34169503
- [Result] Owen N, Healy GN, Matthews CE, Dunstan DW. Too much sitting: the population health science of sedentary behavior. Exerc Sport Sci Rev. 2010 Jul;38(3):105-13. doi: 10.1097/JES.0b013e3181e373a2. PMID 20577058
- [Result] Blodgett J, Theou O, Kirkland S, Andreou P, Rockwood K. The association between sedentary behaviour, moderate-vigorous physical activity and frailty in NHANES cohorts. Maturitas. 2015 Feb;80(2):187-91. doi: 10.1016/j.maturitas.2014.11.010. Epub 2014 Nov 25. PMID 25542406
- [Result] Katzmarzyk PT, Church TS, Craig CL, Bouchard C. Sitting time and mortality from all causes, cardiovascular disease, and cancer. Med Sci Sports Exerc. 2009 May;41(5):998-1005. doi: 10.1249/MSS.0b013e3181930355. PMID 19346988
- [Derived] Rodrigues IB, Kalra M, Zheng R, Rabinovich A, Ioannidis G, Kobsar D, Bray SR, Adachi JD, Fang Q, Papaioannou A. Mapping context of sedentary behaviour in older adults who are prefrail and frail: an analysis of secondary outcomes from a longitudinal study (MAPS-B). BMJ Open. 2024 Nov 27;14(11):e084610. doi: 10.1136/bmjopen-2024-084610. PMID 39609010